CLINICAL TRIAL: NCT01809561
Title: Telomeres Evaluation in Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC13186-12CTIL
Record Dates: First submitted 2013-03-10; First posted 2013-03-12 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-02

CONDITIONS: Endometriosis
Keywords: endometriosis; telomere; telomerase
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples With DNA — whole blood, endometrial tissue biopsy, lesion of endometriosis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- endometriosis: The study group will consist of women with suspected endometriosis facing surgical treatment
  Interventions: Procedure: tissue biopsy during surgical treatment
- no endometriosis: The control group will consist of healthy women facing gynecologic surgery for different indication
  Interventions: Procedure: tissue biopsy during surgical treatment

INTERVENTIONS:
Procedure: tissue biopsy during surgical treatment — The samples collected will test for histological diagnosis of endometriosis and verification tests will be done to characterize the telomeres array and telomerase levels and other characteristics for genomic instability such as spontaneous aneuploidy.
  Other Names: endometriosis tissue biopsy only study group; endometrial tissue biopsy

SUMMARY:
The purpose of the study is to assess the telomere array of different endometriosis tissue and endometrium from women with endometriosis compared to healthy women.

Our hypothesis is that telomere shortening and high telomerase activity will be found in tissues from women with endometriosis.

DETAILED DESCRIPTION:
The purpose of the study is to assess the telomere array of different endometriosis tissue and endometrium from women with endometriosis compared to healthy women. Our hypothesis is that telomere shortening and high telomerase activity will be found in tissues from women with endometriosis, compared to women without endometriosis.

A prospective study that compares telomeres and telomerase levels in different lesions of endometriosis and endometrial tissue of women with endometriosis and healthy women without endometriosis. The study group will consist of women with suspected endometriosis facing surgical treatment and the control group will consist of healthy women facing gynecologic surgery for different indication.

We will sample endometrial tissue in both groups. In the study group we additionally will sample endometriosis lesion.

The samples collected will test for histological diagnosis of endometriosis and verification tests will be done to characterize the telomeres array and telomerase levels and other characteristics for genomic instability such as spontaneous aneuploidy.

expect telomere shortening and high telomerase activity in endometrial tissue and in endometriosis tissue sample, that won't characterize samples from women without endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* women with suspected endometriosis facing surgical treatment

Exclusion Criteria:

* no endometriosis on histology
* malignant finding on histology

Ages: 15 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: women facing surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
characterize the telomeres array and telomerase levels and other characteristics for genomic instability such as spontaneous aneuploidy in endometriosis tissue. | the tissue sample will colect at time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ron Schonman, DR, Study Chair — MeirMc, Israel
Locations (1):
- OBGYN department, Meir Medical Center, Kfar Saba, Israel, Israel

REFERENCES:
- [Background] Sampson JA. Peritoneal endometriosis due to the menstrual dissemination of endometrial tissue into the peritoneal cavity. Am J Obstet Gynecol 1927 14,422-469.
- [Background] Lapp T. ACOG issues recommendations for the management of endometriosis. American College of Obstetricians and Gynecologists. Am Fam Physician. 2000 Sep 15;62(6):1431, 1434. No abstract available. PMID 11011865
- [Background] Wells M. Recent advances in endometriosis with emphasis on pathogenesis, molecular pathology, and neoplastic transformation. Int J Gynecol Pathol. 2004 Oct;23(4):316-20. doi: 10.1097/01.pgp.0000139636.94352.89. PMID 15381900
- [Background] Sharpe-Timms KL. Endometrial anomalies in women with endometriosis. Ann N Y Acad Sci. 2001 Sep;943:131-47. doi: 10.1111/j.1749-6632.2001.tb03797.x. PMID 11594534
- [Background] Nolan CM. Human immunodeficiency syndrome-associated tuberculosis: a review with an emphasis on infection control issues. Am J Infect Control. 1992 Feb;20(1):30-4. doi: 10.1016/s0196-6553(05)80123-3. No abstract available. PMID 1554145
- [Background] Jones RK, Searle RF, Bulmer JN. Apoptosis and bcl-2 expression in normal human endometrium, endometriosis and adenomyosis. Hum Reprod. 1998 Dec;13(12):3496-502. doi: 10.1093/humrep/13.12.3496. PMID 9886539
- [Background] Meresman GF, Vighi S, Buquet RA, Contreras-Ortiz O, Tesone M, Rumi LS. Apoptosis and expression of Bcl-2 and Bax in eutopic endometrium from women with endometriosis. Fertil Steril. 2000 Oct;74(4):760-6. doi: 10.1016/s0015-0282(00)01522-3. PMID 11020520
- [Background] Higashiura Y, Kajihara H, Shigetomi H, Kobayashi H. Identification of multiple pathways involved in the malignant transformation of endometriosis (Review). Oncol Lett. 2012 Jul;4(1):3-9. doi: 10.3892/ol.2012.690. Epub 2012 Apr 23. PMID 22807950
- [Background] Amiel A, Gronich N, Yukla M, Suliman S, Josef G, Gaber E, Drori G, Fejgin MD, Lishner M. Random aneuploidy in neoplastic and pre-neoplastic diseases, multiple myeloma, and monoclonal gammopathy. Cancer Genet Cytogenet. 2005 Oct 1;162(1):78-81. doi: 10.1016/j.cancergencyto.2005.03.006. PMID 16157205
- [Background] Amiel A, Yukla M, Gaber E, Leopold L, Josef G, Fejgin M, Lishner M. Random aneuploidy in CML patients at diagnosis and under imatinib treatment. Cancer Genet Cytogenet. 2006 Jul 15;168(2):120-3. doi: 10.1016/j.cancergencyto.2006.02.002. PMID 16843101
- [Background] Saini N, Srinivasan R, Chawla Y, Sharma S, Chakraborti A, Rajwanshi A. Telomerase activity, telomere length and human telomerase reverse transcriptase expression in hepatocellular carcinoma is independent of hepatitis virus status. Liver Int. 2009 Sep;29(8):1162-70. doi: 10.1111/j.1478-3231.2009.02082.x. Epub 2009 Jul 17. PMID 19627485
- [Background] Svenson U, Roos G. Telomere length as a biological marker in malignancy. Biochim Biophys Acta. 2009 Apr;1792(4):317-23. doi: 10.1016/j.bbadis.2009.01.017. Epub 2009 Feb 7. PMID 19419696
- [Background] Yokoyama Y, Takahashi Y, Morishita S, Hashimoto M, Niwa K, Tamaya T. Telomerase activity in the human endometrium throughout the menstrual cycle. Mol Hum Reprod. 1998 Feb;4(2):173-7. doi: 10.1093/molehr/4.2.173. PMID 9542976
- [Background] Lehner R, Enomoto T, McGregor JA, Shroyer AL, Haugen BR, Pugazhenthi U, Shroyer KR. Quantitative analysis of telomerase hTERT mRNA and telomerase activity in endometrioid adenocarcinoma and in normal endometrium. Gynecol Oncol. 2002 Jan;84(1):120-5. doi: 10.1006/gyno.2001.6474. PMID 11748987
- [Background] Kim CM, Oh YJ, Cho SH, Chung DJ, Hwang JY, Park KH, Cho DJ, Choi YM, Lee BS. Increased telomerase activity and human telomerase reverse transcriptase mRNA expression in the endometrium of patients with endometriosis. Hum Reprod. 2007 Mar;22(3):843-9. doi: 10.1093/humrep/del425. Epub 2006 Oct 31. PMID 17077107
- [Background] Hapangama DK, Turner MA, Drury JA, Quenby S, Saretzki G, Martin-Ruiz C, Von Zglinicki T. Endometriosis is associated with aberrant endometrial expression of telomerase and increased telomere length. Hum Reprod. 2008 Jul;23(7):1511-9. doi: 10.1093/humrep/den172. Epub 2008 May 2. PMID 18456668
- [Background] Halme J, Hammond MG, Hulka JF, Raj SG, Talbert LM. Retrograde menstruation in healthy women and in patients with endometriosis. Obstet Gynecol. 1984 Aug;64(2):151-4. PMID 6234483